CLINICAL TRIAL: NCT05237596
Title: Erosive Osteoarthritis of the Hand: Efficacy of Prescription-grade Crystalline Glucosamine Sulfate as an add-on Therapy to Conventional Treatments
Brief Title: Prescription-grade Crystalline Glucosamine Sulfate Therapy in Erosive Hand Osteoarthritis
Status: Completed | Type: Observational
Sponsor: University of Siena (Other)
Responsible Party: Principal Investigator, fioravanti antonella, Principal Investigator, University of Siena
Other Study IDs: pCGS_EHOA
Record Dates: First submitted 2022-02-02; First posted 2022-02-14 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Erosive Osteoarthritis of the Hand
MeSH Terms: interventions — Glucosamine; Acetaminophen

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Prescription-grade Crystalline Glucosamine Sulfate Group (pCGS Group): pCGS Group includes patients treated with pCGS (Dona®, VIATRIS), in sachets of powder for oral solution, at the dose of 1500 mg glucosamine sulfate once daily, for a total period of 6 consecutive months according to the approved indication for knee OA, in addition to conventional therapy for HOA.
  Interventions: Drug: Glucosamine Sulfate
- Control Group: Control Group includes patients treated with conventional therapy alone for at least 6 consecutive months.

INTERVENTIONS:
Drug: Glucosamine Sulfate — Treatment for at least 6 months with prescription-grade crystalline Glucosamine Sulfate in addition to conventional treatment
  Other Names: Acetaminophen; Non-steroidal anti-inflammatory drugs
  Groups: Prescription-grade Crystalline Glucosamine Sulfate Group (pCGS Group)

SUMMARY:
The objective of this study is to evaluate the efficacy of prescription-grade Crystalline Glucosamine Sulfate (pCGS), as an add-on treatment to conventional therapy, compared to usual therapy alone, in patients with erosive osteoarthritis of the hand (EHOA).

This is a 6-months retrospective study including patients with concomitant gonarthrosis and EHOA, defined as the presence of central erosion in at least two interphalangeal joints. Eligibility criteria are symptoms duration for at least 3 months, with a global hand pain score ≥40 mm on a 0-100 Visual Analogue Scale (VAS) and a Functional Index for Hand Osteoarthritis (FIHOA) score ≥6. The participants are stratified into two groups based on whether or not pCGS, at the daily dose of 1500 mg, was added to the conventional therapy for hand osteoarthritis (HOA). The latter consists of education and training in ergonomic principles, exercise and the use on-demand of acetaminophen or oral non-steroidal anti-inflammatory drugs. Patients are evaluated at baseline, after 3 and 6 months. Primary outcome measures are the change from baseline to month 6 in VAS and in FIHOA score. Secondary outcomes are duration of morning stiffness, health assessment questionnaire (HAQ), medical outcomes study 36-item short form (SF-36), symptomatic drugs consumption and percentage of treatment responders, according to the OMERACT/OARSI criteria.

ELIGIBILITY:
Inclusion Criteria:

* Erosive Hand Osteoarthritis, defined as the presence of the classical central erosion in at least two interphalangeal joints
* Treatment for at least 6 consecutive months with prescription-grade crystalline GS at the daily dose of 1500 mg in addition to the conventional therapy or with usual care alone.
* Symptoms duration for at least 3 months defined as global hand pain score superior to 40 mm on a 0-100 VAS and a FIHOA score of at least 6.

Exclusion Criteria:

* Medical history of any inflammatory joint disease, septic arthritis, previous articular fracture of the concerned joints, or the presence of any other rheumatic diseases that could cause secondary OA, such as hemochromatosis
* Concomitant therapy with SYSADOAs, other than pCGS, steroids by any route of administration and intra-articular injection of any joint with hyaluronic acid during the previous 6 months
* Concomitant treatment with intra-muscular or intra-venous bisphosphonates in the previous 6 months
* Contraindications or special warnings for pCGS presented in the data sheet.

Ages: 48 Years to 87 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants are stratified into two groups (pCGS Group and Control Group) based on whether or not prescription-grade crystalline GS treatment, prescribed for the actually approved indication of knee OA, was added to the conventional therapy. This stratification is based on regrouping patients with similar clinical characteristics at baseline.
Sampling Method: Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2021-01-07 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Difference between the two groups in the change of the patient's assessment of global hand pain on a 0- 100 mm Visual Analogue Scale | Basal time; three months; six months
  0-100 mm scale with 0 representing the absence of pain
Difference between the two groups in the change of the Functional Index for Hand Osteoarthritis (FIHOA) score | Basal time; three months; six months
  The FIHOA score represents a quantitative measure of functional disability of the hands; it contains 10 items and is an investigator-administered questionnaire. Patients are asked to answer each item using a four-point Likert scale: 0 = possible without difficulty, 1 = possible with slight difficulty, 2 = possible with considerable difficulty, 3 = impossible; the range of scores is 0-30 and the highest values indicate the worst functionality. The validate Italian version of FIHOA is used for the present study

SECONDARY OUTCOMES:
Difference between the two groups in the change in the duration of morning stiffness | Basal time; three months; six months
  VAS stiffness is measured in minutes and based on the self-report of patients
Difference between the two groups in the change of HAQ | Basal time; three months; six months
  HAQ is a self administered questionnaire developed to measure disability consisting of 8 sections: dressing arising, eating, walking, hygiene, reach, grip, and activities and ranging from 0 to 3 with a higher score corresponding to worse disability
Difference between the two groups in the change of SF-36 | Basal time; three months; six months
  SF-36 is a widely used measure of health and wellbeing, including two main domains, mental and physical component summary (MCS and PCS respectively), that investigates 8 different areas of perceived health, such as physical functioning, physical role, bodily pain, general health, vitality, social functioning, emotional role and mental health. Scores range from "0 to 100" where "0" indicates the worst condition and "100" indicates the best possible condition
NSAIDs and/or acetaminophen consumption | Basal time; three months; six months
  The acetaminophen and NSAIDs/COX-2 inhibitors consumption was calculated asking the patients at each visit the number of tablets taken weekly.
OMERACT/OARSI criteria responders | Basal time; three months; six months
  percentage of treatment responders at 3 and 6 months, according to the Outcome Measures in Rheumatology (OMERACT) and Osteoarthritis Research Society International (OARSI) criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Rheumatology Unit Azienda Ospedaliera Universitaria Senese, Siena, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tenti S, Veronese N, Cheleschi S, Seccafico I, Bruyere O, Reginster JY, Fioravanti A. Prescription-grade crystalline glucosamine sulfate as an add-on therapy to conventional treatments in erosive osteoarthritis of the hand: results from a 6-month observational retrospective study. Aging Clin Exp Res. 2022 Jul;34(7):1613-1625. doi: 10.1007/s40520-022-02151-7. Epub 2022 May 30. PMID 35637324